CLINICAL TRIAL: NCT00415298
Title: AP5346 for Recurrent/Unresectable Squamous Cell Carcinoma of the Head and Neck: A Pilot Study With Clinical and Biological Endpoints
Brief Title: AP5346 or Oxaliplatin in Treating Patients With Metastatic and/or Unresectable Recurrent Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000520463; UCSD-HRPP-050275
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2007-05

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — ProLindac; Oxaliplatin; Gene Expression Profiling; Immunohistochemistry; Biopsy

INTERVENTIONS:
Drug: DACH polymer platinate AP5346
Drug: oxaliplatin
Genetic: gene expression analysis
Other: immunohistochemistry staining method
Other: pharmacological study
Procedure: biopsy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as AP5346 and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This randomized clinical trial is studying the dose of AP5346 to see how well it works compared with the dose of oxaliplatin in treating patients with metastatic and/or unresectable recurrent head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the delivered-dose of platinum per gram of wet weight from a single dose of AP5346 vs a single dose of oxaliplatin in patients with metastatic and/or unresectable recurrent squamous cell carcinoma of the head and neck (SCCHN).
* Correlate platinum accumulation in the tumor and tumor DNA with clinical response in patients treated with these regimens.
* Correlate platinum accumulation in the tumor and tumor DNA with molecular tumor response as determined by GADD153 expression in patients treated with these regimens.
* Quantify, by immunohistochemistry, the expression of the copper transporters CTR1, ATP7A, and ATP7B in SCCHN tumors and correlate expression of these transporters with tumor platinum levels.
* Determine response in patients treated with AP5346.
* Obtain additional data on the safety of AP5346 in these patients.

OUTLINE: This is a randomized, pilot study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive AP5346 IV over 2 hours three times daily on days 1 and 15.
* Arm II: Patients receive a single dose of unmodified oxaliplatin IV over 2 hours on day 1.

Beginning on day 29, all patients may receive AP5346 as in arm I. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor biopsy before and 24 hours after the first course of treatment for correlative pharmacological, immunohistochemical (IHC), and molecular studies. Tumor specimens are assessed for platinum content, GADD153 gene expression (by molecular analysis), and copper transporter (CTR1, ATP7A, ATP7B) expression by IHC.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary squamous cell carcinoma of the head and neck, including the oral cavity, oropharynx, hypopharynx, larynx, or nasopharynx

  * Metastatic and/or unresectable locally recurrent disease for which no curative treatment is available

    * Patients must not be candidates for surgical resection or radiotherapy with curative intent
    * Histological documentation of relapse required, especially for locoregional recurrence or recurrence in a previously irradiated field
* Tumor(s) must be amenable to minimally invasive biopsy during the first course of treatment

  * Must have evidence of progression or appearance of a new lesion after completion of radiotherapy, if biopsy site is in a previously irradiated field

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Absolute neutrophil count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Bilirubin < 1.5 times upper level of normal (ULN)
* Alkaline phosphatase (AP) ≤ 5 times normal (unless elevation is due to bone disease or bone metastasis in the absence of liver disease)
* AST and ALT ≤ 3 times ULN

  * AST and ALT > 3 times ULN allowed provided AP ≤ 3 times ULN
* Blood urea < 1.5 times ULN
* Creatinine < 1.5 times ULN OR creatinine clearance > 60 mL/min OR creatinine clearance by 24-hour urine collection normal
* Calcium normal
* No history of hypersensitivity reactions of any kind to cisplatin or carboplatin
* No other serious medical condition or psychiatric illness that would preclude the patient's ability to give informed consent or receive study treatment
* No symptomatic peripheral neuropathy ≥ grade 2
* No need for IV alimentation
* No other serious illness or medical condition, including, but not limited to, the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris or cardiac arrhythmia
  * Significant neurologic or psychiatric disorders, including dementia or uncontrolled seizures
  * Hypophosphatemia

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior and no other concurrent anticancer treatment (i.e., chemotherapy, chemoradiotherapy, or radiotherapy)
* At least 4 weeks since prior biologic therapy
* No prior oxaliplatin

  * Prior cisplatin or carboplatin allowed
* No concurrent anticoagulants other than cardioprotective doses of aspirin, cyclooxygenase 1-inhibitory nonspecific anti-inflammatory drugs, or prophylactic low-dose heparin
* Concurrent bisphosphonates for hypercalcemia allowed provided the drug was initiated ≥ 3 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-05

PRIMARY OUTCOMES:
Delivered-dose of platinum 24 hours after IV injection of a single dose of AP5346 vs a single dose of oxaliplatin
Correlation of platinum accumulation in the tumor and tumor DNA with clinical response
Correlation of platinum accumulation in the tumor and tumor DNA with molecular response as determined by GADD153 expression
Quantification of expression of CTR1, ATP7A, and ATP7B in squamous cell carcinoma of the head and neck (SCCHN) tumors by immunohistochemistry
Correlation of expression of CTR1, ATP7A, and ATP7B in SCCHN tumors with tumor platinum levels
Toxicity of AP5346

CONTACTS AND LOCATIONS:
Overall Officials: William L. Read, MD, Study Chair — University of California, San Diego
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States